CLINICAL TRIAL: NCT04817501
Title: Phenotypic Spectrum of Circulating Tumor Cell Populations as Markers of Liquid Biopsy in Tumors of the Female Reproductive System
Brief Title: Phenotypic Spectrum of CTCs in Tumors of the Female Reproductive System
Acronym: CTCs
Status: Completed | Type: Observational
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: CTC Phenotyping
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer; Ovarian Cancer; Endometrial Cancer
Keywords: breast cancer; endometrial Cancer; ovarian cancer; CTC heterogeneity; cancer stem cells; epithelial-mesenchymal transition; multicolor flow cytometry; liquid biopsy; circulating tumor cell
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA-stabilized venous blood (5 mL) EDTA-stabilized ascitic fluid (5 mL)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Breast cancer: At least eighty five subjects with breast cancer
  Interventions: Other: Taking 5 ml of venous blood at different time intervals; Other: Taking 5 ml EDTA-stabilized ascitic fluid sampled during laparoscopy if any
- Ovarian cancer: At least 32 subjects with ovarian cancer
  Interventions: Other: Taking 5 ml of venous blood at different time intervals; Other: Taking 5 ml EDTA-stabilized ascitic fluid sampled during laparoscopy if any
- Endometrial Cancer: At least 33 subjects with endometrial cancer
  Interventions: Other: Taking 5 ml of venous blood at different time intervals; Other: Taking 5 ml EDTA-stabilized ascitic fluid sampled during laparoscopy if any
- Healthy control: 30 healthy volunteers
  Interventions: Other: Taking 5 ml of venous blood at different time intervals
- Suspected malignant tumor non-verified: Patients with suspected malignant tumor, which was not verified by biopsy. Nubmber of patients to be defined
  Interventions: Other: Taking 5 ml of venous blood at different time intervals; Other: Taking 5 ml EDTA-stabilized ascitic fluid sampled during laparoscopy if any

INTERVENTIONS:
Other: Taking 5 ml of venous blood at different time intervals
  Other Names: Taking 5 ml EDTA-stabilized ascitic fluid sampled during laparoscopy
Other: Taking 5 ml EDTA-stabilized ascitic fluid sampled during laparoscopy if any
  Groups: Breast cancer; Endometrial Cancer; Ovarian cancer; Suspected malignant tumor non-verified

SUMMARY:
The study evaluates the level and molecular profiles of different CTC populations as markers for predicting the risk of developing hematogenous metastases and the effectiveness of treatment in patients with tumors of the female reproductive system (breast cancer, endometrial cancer, and ovarian cancer).

The primary objective are:

1. To assess the presence and number of different populations of CTCs at different time points (before biopsy, before surgery, and after surgery).
2. To assess the relationships of different CTCs populations prior to treatment initiation with the effects of neoadjuvant chemotherapy and the risks of recurrence and metastases.
3. To assess the molecular profiles of different CTCs populations in the blood and in ascitic fluid.

The secondary objective is to compare the multicolor flow cytometry results with data of ultrasound, CT and/or MRI, serum tumor markers, and immunohistochemical studies in patients with breast cancer, endometrial cancer and ovarian cancer

DETAILED DESCRIPTION:
The overall goal is to study the diagnostic and prognostic efficacy of various CTC populations as liquid biopsy markers in tumors of the female reproductive system (breast cancer, endometrial cancer, and ovarian cancer).

Phase I study:

Determination of different populations of CTCs in blood and ascitic fluid (if any) prior to treatment.

The main objectives of the study:

1. To assess the presence and number of different CTC populations at different time points (before biopsy and before surgery) using multicolor flow cytometry.
2. To assess the relationships between different CTCs populations prior to treatment initiation with the effects of neoadjuvant chemotherapy and the risks of recurrence and metastases.
3. To assess the molecular profiles of different CTCs populations in the blood and in ascitic fluid.

Additional research tasks:

To compare the multicolor flow cytometry results with the data of ultrasound, CT and/or MRI, serum tumor markers, and immunohistochemical studies in patients with breast cancer, endometrial cancer, and ovarian cancer Methodology: Open-label, exploratory, single centre study. Blood and ascitic fluid collected from subjects (if available)

ELIGIBILITY:
Inclusion Criteria:

* Subject is > 18 years of age A negative pregnancy test (serum beta-human chorionic gonadotropin, beta-HCG) at screening for all patients of childbearing potential.
* Clinical and radiological diagnosis of breast cancer or Ovarian cancer or Endometrial Cancer General satisfactory condition (according to the ECOG scale ≤2) Subject is capable to undergo the diagnostic investigations to be performed in the study
* Informed consent

Exclusion Criteria:

* Active current autoimmune disease or history of autoimmune disease

  * Active infection or history of severe infection within the previous 3 months (if clinically relevant at screening)
  * Known HIV positive or chronically active hepatitis B or C The subject has multiple primary malignant tumors

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender Based: women for breast cancer, Ovarian cancer, Endometrial Cancer
Study Population: Women over 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-02-14 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
CTC phenotype | 6 hours
  Different populations of CTCs are evaluated by multicolor flow cytometry and may include:
  СTC, ascitic tumor cells with stemness features without EMT features; CTC, ascitic tumor cells without stemness and EMT features; CTC, ascitic tumor cells without stemness features and with EMT features; CTC, ascitic tumor cells with stemness features and EMT features; Atypical/hybrid cells without stemness features; Atypical cells.

CONTACTS AND LOCATIONS:
Overall Officials: Evgeniya Kaigorodova, Principal Investigator — Tomsk NRMC
Locations (1):
- Evgeniya Kaigorodova, Tomsk, Tomsk Oblast, Russia